CLINICAL TRIAL: NCT01043107
Title: Study on the Relationship Between The Computer Radiation and The Recrudesce Rate of Thyroid Cancer
Brief Title: Relationship Between Computer and Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Yilong Wu, GGH
Other Study IDs: CancerRe-008; 83827218 (Other: GGH)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-01

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Compuer radiaton group
- control group

SUMMARY:
Thyroid Cancer is one of the most common malignant carcinomas. The incidence of thyroid cancer has risen in the past years. The recrudesce rate is highly raised. Computer is widely used by people nowadays, is it a predisposing factor to the highly raised recrudesce rate? This research observed two random assigned groups, in which the patients were diagnosed by pathologic results. One group were strictly prohibit with using computer, the other were not told. Finally collect the recrudesce rate of each group, analyze the data by statistic software.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid cancer

Exclusion Criteria:

* Non-Thyroid cancer

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population of city of Guangdong province
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-02

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China